CLINICAL TRIAL: NCT00143117
Title: A Phase 2b, Multi-Center, Double-Blind, Placebo-Controlled, Parallel Group Dose Response Study to Assess the Efficacy and Safety of Oral UK-390,957 in Men With Premature Ejaculation
Brief Title: Assessment of Efficacy and Safety of UK-390,957 in Men With Premature Ejaculation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3871022
Record Dates: First submitted 2005-08-30; First posted 2005-09-02 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Ejaculation

INTERVENTIONS:
Drug: UK-390,957

SUMMARY:
To determine whether UK-390,957 is an effective and safe treatment for premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* Premature ejaculation as defined by DSM-IV

Exclusion Criteria:

* History of erectile dysfunction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460
Dates: Start 2004-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy and safety

SECONDARY OUTCOMES:
Assessment of Quality of Sexual Life

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (51):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Atherton, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Laguna Woods, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Redwood City, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Tarzana, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Michigan City, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Saint Clair Shores, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Southhaven, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Edison, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Voorhees Township, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3871022&StudyName=Assessment+of+Efficacy+and+Safety+of+UK%2D390%2C957+in+Men+With+Premature+Ejaculation